CLINICAL TRIAL: NCT07189442
Title: Combining L-theanine and Paraxanthine for Transient Improvement of Cognitive Deficits Among Patients With Attention Deficit Hyperactivity Disorder and Autism Spectrum Disorder: A Series of Translational Pilot Neuroimaging Studies
Brief Title: L-theanine and Paraxanthine for Cognitive Improvement in Adults With ADHD and ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Principal Investigator, Samudani Dhanasekara, Assistant Professor, Texas Tech University Health Sciences Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB2025-147
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Autism Spectrum Disorder (ASD)
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; ASD; Autism spectrum disorder; Autism
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Autistic Disorder | interventions — theanine; 1,7-dimethylxanthine

STUDY DESIGN:
Intervention Model Description: Crossover Assignment (two-way, repeated measures)
Who Masked: Participant
Masking Description: Single (Participant and outcomes assessors blinded; study staff preparing capsules unblinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention deficit hyperactivity disorder (ADHD) (Experimental): A group of 12 adult males with Attention Deficit Hyperactivity Disorder (ADHD) will be enrolled. Each participant will receive both study conditions in a randomized, single-blinded, repeated-measures crossover design:
  Active Condition: One capsule containing 200 mg L-theanine + 200 mg paraxanthine.
  Placebo Condition: One capsule containing 400 mg of corn starch. The order of administration will be randomized, with each participant completing both conditions on separate visits (visits 2 and 3).
  Interventions: Dietary Supplement: L-theanine and paraxanthine; Dietary Supplement: Placebo
- Autism spectrum disorder (ASD) (Experimental): A group of 12 adult males with autism spectrum disorder (ASD) will be enrolled. Each participant will receive both study conditions in a randomized, single-blinded, repeated-measures crossover design:
  Active Condition: One capsule containing 200 mg L-theanine + 200 mg paraxanthine.
  Placebo Condition: One capsule containing 400 mg of corn starch. The order of administration will be randomized, with each participant completing both conditions on separate visits (visits 2 and 3).
  Interventions: Dietary Supplement: L-theanine and paraxanthine; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-theanine and paraxanthine — 200 mg L-theanine + 200 mg paraxanthine capsule
Dietary Supplement: Placebo — 400 mg corn starch capsule

SUMMARY:
This pilot study will test whether combining L-theanine and paraxanthine improves sustained attention, inhibitory control, and overall cognition in adults with ADHD and ASD. Two parallel randomized, single-blinded, repeated-measures crossover trials will be conducted. Participants will complete neuropsychological testing, fMRI scanning, and self-report measures following administration of the L-theanine-paraxanthine combination compared to placebo.

DETAILED DESCRIPTION:
Improving cognitive functions, including how fast the brain processes information, staying focused, and controlling impulsive actions, has been a topic of interest for centuries. These functions are frequently impaired in developmental or neurological conditions like attention-deficit hyperactivity disorder (ADHD) and autism spectrum disorder (ASD). Although medications like amphetamines can help manage cognitive deficits, they often carry significant side effects, risk of addiction, and high costs. Consequently, many individuals and families turn to complementary and alternative treatments. For instance, people with neurodevelopmental conditions, including ADHD, may consume more caffeinated beverages in the hope of boosting cognitive performance. This highlights the need for the exploration of commonly available alternative approaches to determine their efficacy. This study specifically aims to investigate an alternative approach that could serve as a more affordable, integrative, and complementary treatment modality for ADHD and ASD.

Findings of recent controlled cognitive and fMRI studies corroborate the findings of others to indicate that intake of two constituents of tea and coffee, namely L-theanine and caffeine, improves sustained attention in healthy young adult males by decreasing mind wandering. Interestingly, when administered together, L-theanine and caffeine synergistically acted to reduce mind wandering while engaged in a cognitively demanding task. Given the low cost and safety, oral administration of the L-theanine-caffeine combination seems to be a promising strategy to alleviate ADHD-associated impairments of sustained attention. However, regular high consumption of caffeine has adverse effects, such as jitteriness and sleep disturbance due to its metabolites, and the metabolism of caffeine has individual variability.

Paraxanthine is an active metabolite of caffeine that has cognitive benefits without adverse effects and predictable metabolism. However, the effects of the L-theanine-paraxanthine combination on improving cognitive deficits of adults with ADHD and ASD have not been examined. It is expected that combining theanine with paraxanthine instead of caffeine would result in more predictable, consistent, and possibly more marked improvements. There is a critical need to establish the efficacy and mechanisms of action of the L-theanine-paraxanthine combination in order to improve ADHD and ASD-related cognitive deficits. Therefore, the investigators plan to conduct a randomized, single-blinded, repeated-measures crossover trial to answer the following research questions.

ELIGIBILITY:
Inclusion Criteria:

Adults (18+ years) diagnosed by a physician (per self-report) with ADHD or ASD

* Participants with a dual diagnosis and ASD and ADHD will be recruited but will only be included in the ASD group - their concurrent ADHD diagnosis will be included as an additional variable in exploratory analyses

Exclusion Criteria:

1. Subjects with gross visual or auditory impairments that might limit their ability to perform neuropsychological tasks
2. Inability to read and follow written instructions
3. Physical, neurological, intellectual, or psychiatric impairments (except ADHD or ASD) that could affect cognitive and motor functions
4. Subjects on medications including antidepressants and antipsychotics that may affect performance in the tasks
5. Subjects on medications that are likely to interact with the administered substances, including regular intake of medication that could alter visual, auditory, cognitive, or motor functions (except stimulants)
6. History of head injury resulting in loss of consciousness/history of brain surgery
7. Subjects who have developed adverse effects when caffeine/paraxanthine /L-theanine/corn starch (will be in placebo) containing products were consumed
8. Subjects who are unwilling or unable to refrain from intake of L-theanine/ caffeine/ paraxanthine containing food or beverages within the 24 hours prior to each study visit
9. Intake of drugs containing caffeine, other phosphodiesterase inhibitors, or adenosine receptor blockers within the past 3 months
10. Intake of medications known to have pharmacological interactions with paraxanthine within the past 3 months
11. Current/past diagnosis of tics or other forms of dyskinesia
12. History of headache, drowsiness, anxiety, insomnia, or nausea following intake of caffeine or caffeine-containing beverages
13. Current/past history of smoking and/or alcohol or drug abuse
14. Subjects with absolute contraindications to undergo MRI after being screened by the TTNI safety screening sheet (Appendix)
15. Unwillingness or inability to entirely refrain from the use of electronic devices during study visits
16. Unwillingness or inability to follow written, on-screen, and verbal instructions given by the study team.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
fMRI task-related activity | At visit 2 or 3, 30 minutes after intake of L-theanine-paraxanthine or placebo.
  fMRI task-related activity in default mode and central executive networks during Go/NoGo and Stop-Signal tasks.
Stop Signal Reaction Time | At visit 2 or 3, 30 minutes after intake of L-theanine-paraxanthine or placebo. This task is performed while in the MRI.
  Estimated time (milliseconds) required to inhibit a prepotent response following a stop signal, computed using the horse-race model and drift-diffusion theory. Lower values indicate better inhibitory control.
d-prime (sensitivity to the Go signal) | At visit 2 or 3, 30 minutes after intake of L-theanine-paraxanthine or placebo. This task is performed while in the MRI.
  d-prime on Go/No-Go task computed using the signal detection theory.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data may be shared with qualified researchers upon a reasonable request and after obtaining institutional approval.